CLINICAL TRIAL: NCT01803321
Title: A Pilot, Multi-center, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose, Safety, Tolerability and Preliminary Efficacy Study of Two Dose Levels of IL-1 Trap Administered Subcutaneously in Pediatric Subjects With Active Systemic Juvenile Idiopathic Arthritis (SJIA)
Brief Title: Study to Evaluate the Safety and Tolerability of Two Doses of Rilonacept in Pediatric Subjects With Active Systemic Juvenile Idiopathic Arthritis (SJIA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IL1T-AI-0504
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
Keywords: SJIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Dose 1
  Interventions: Drug: rilonacept (IL-1 Trap); Other: Placebo
- Cohort 2 (Experimental): Dose 2
  Interventions: Drug: rilonacept (IL-1 Trap); Other: Placebo

INTERVENTIONS:
Drug: rilonacept (IL-1 Trap)
Other: Placebo

SUMMARY:
This study is a pilot, ascending dose, multi-center, randomized, double blind, placebo controlled, pediatric study conducted in three phases.

ELIGIBILITY:
Inclusion Criteria include, but are not limited to, the following:

* Patients aged 4 to less than 21 years who meet the criteria for active SJIA
* Must have been on a stable dose of non-steroidal anti-inflammatory drugs (NSAIDs) for at least 4 weeks prior to the screening visit

Exclusion Criteria include, but are not limited to, the following:

* Use of certain medications prior to the baseline visit
* History of recurrent infections

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events (TEAEs) | Baseline to Week 123

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (9):
- United States (9):
  - Los Angeles, California
  - Wilmington, Delaware
  - Chicago, Illinois
  - Hackensack, New Jersey
  - Long Island City, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dallas, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Lovell DJ, Giannini EH, Reiff AO, Kimura Y, Li S, Hashkes PJ, Wallace CA, Onel KB, Foell D, Wu R, Biedermann S, Hamilton JD, Radin AR. Long-term safety and efficacy of rilonacept in patients with systemic juvenile idiopathic arthritis. Arthritis Rheum. 2013 Sep;65(9):2486-96. doi: 10.1002/art.38042. PMID 23754188